CLINICAL TRIAL: NCT07211204
Title: Study To Compare The Efficacy Of Cervical Cytology With Molecular Screening In The Detection Of Reactive Cellular Changes In The Cervix In An Open Population
Brief Title: Comparison Of Cytology And Molecular Screening For Detecting Cervical Reactive Cellular Changes In General Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Timser SAPI de CV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: PROT-ATSO-INV-003; 2024-EXT-886 (Other: Ethics Committee of Medica Sur)
Record Dates: First submitted 2025-06-03; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Atypical Squamous Cell of Undetermined Significance; ASC-US; Atypical Glandular Cells of Uncertain Significance; AGUS; Cervical Intraepithelial Neoplasia (CIN); CIN 1; CIN 2; CIN 3; Cervical Cancer
Keywords: Cervical precursor lesions; Reactive cellular changes; Cervical cancer
MeSH Terms: conditions — Atypical Squamous Cells of the Cervix; Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — Restraint, Physical; Human Papillomavirus DNA Tests; Colposcopy; Biopsy

STUDY DESIGN:
Intervention Model Description: Group 1. All participants will receive a colposcopy, Pap smear, and a venipuncture. Diagnosis by colposcopy will set four clinical groups: negative control (CTR), low-grade squamous intraepithelial lesions LSIL (CIN-1), high-grade squamous intraepithelial lesions HSIL (CIN-2/3), and cervical cancer (CC).
  Group 2. The participants in groups LSIL, HSIL, and CC will be biopsied. The histopathology analysis of the biopsy is the gold standard for the diagnosis.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Given this is a screening study:
  I) Participant. All enrolled participants will be asymptomatic women. Group assignment will be defined after colposcopy or histopathology (when applicable).
  II) Care Provider. The gynecologist will not have a priori knowledge of the condition of the participant. During colposcopy only those participants with abnormal results will be biopsied.
  III) Investigator. None of the investigators performing the tests (cytology, HPV detection, molecular screening, or histopathology) will know each other's results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Screening for reactive cellular changes in the cervix (Other): Participants will be drawn from an open population, so they will be asymptomatic for any cervical disease. Based on colposcopy, there will be four clinical groups: negative control (CTR), low-grade squamous intraepithelial lesion (LSIL, CIN-1), high-grade squamous intraepithelial lesion (HSIL, CIN-2/3), and cervical cancer (CC).
  Interventions: Procedure: Physical examination; Other: Liquid-based cytology; Other: Molecular screening; Other: HPV DNA test; Diagnostic Test: Colposcopy
- Histopathology of cervical biopsy (Other): Based on colposcopy, participants in the groups LSIL/CIN-1, HSIL/CIN-2/3, and cervical cancer (CC) will be biopsied.
  Interventions: Diagnostic Test: Histopathology

INTERVENTIONS:
Procedure: Physical examination — Physical examination and interview for obtaining a medical record
  Other Names: Clinical examination
  Arms: Screening for reactive cellular changes in the cervix
Other: Liquid-based cytology — Screening test for cervical precursor lesions and/or cancer. LBC is a procedure in which a cervical smear is examined under the microscope.
  Other Names: LBC
  Arms: Screening for reactive cellular changes in the cervix
Other: Molecular screening — The molecular screening detects three human biomarkers associated with cervical precursor lesions and/or cervical cancer. Biomarker detection is done by Western blot and ELISA in human sera.
  Other Names: Circulating biomarker screening
  Arms: Screening for reactive cellular changes in the cervix
Other: HPV DNA test — HPV DNA detection is performed using a cervical swab.
  Other Names: HPV PCR test; HPV screening; HPV detection; Human papillomavirus DNA test
  Arms: Screening for reactive cellular changes in the cervix
Diagnostic Test: Colposcopy — A diagnostic procedure to visually examine the cervix, vagina, and vulva with a colposcope.
  Arms: Screening for reactive cellular changes in the cervix
Diagnostic Test: Histopathology — Is the definitive diagnosis of cervical precursor lesions and cervical cancer. It is the microscopic study of diseased cells and tissues stained with hematoxylin and eosin.
  Other Names: Cervical biopsy; Biopsy; Histopathologic examination; Histopathologic analysis; Hematoxylin and eosin stain (H&E) in histopathology
  Arms: Histopathology of cervical biopsy

SUMMARY:
This study compares the efficacy of cytology (Pap smear) with the molecular screening in their ability to detect reactive cellular changes in the cervix among an open population

DETAILED DESCRIPTION:
The primary goal of this study is to compare the efficacy of the cytology (Pap smear) with the molecular screening -of three human biomarkers- in their ability to detect reactive cellular changes in the cervix among an open population. Participants will be asked to attend two study visits. All the clinical procedures will be done on the first visit:

1. Explanation of the study and its procedures. Only participants that give their written Informed Consent will be enrolled in the study.
2. Interview and physical examination to obtain a medical record. The interview will collect information related to known risks factors for cervical lesions.
3. Venipuncture to obtain a blood sample.
4. Colposcopy to obtain a cervical smear and a colposcopic diagnosis. The cervical smear will be used to perform liquid-based cytology and HPV detection.
5. Biopsy, only if the gynecologist detects a cervical lesion or another abnormality during colposcopy.

The gynecologist will make preliminary recommendations based on the colposcopic findings.

During the second visit the study's gynecologist will explain the tests' results and provide clinical recommendations to each participant.

The sensitivity, specificity, and predictive values of cytology, HPV detection, and molecular screening will be calculated using colposcopy (for all participants) and histopathology (for those biopsied). These results will be compared using a DeLong test. Correlation tests will be performed using risk factors data and test results.

ELIGIBILITY:
Inclusion Criteria:

* Be in good general health.
* Age 18-85 years.
* A minimum fast of 6 hours and no more than 12 hours.
* Refrain from sexual intercourse 24 hours before the study.
* Give written informed consent.

Exclusion Criteria:

* Having a subtotal, total, or radical hysterectomy.
* Being pregnant or suspected of being pregnant. A rapid urine test will be performed. If the result is positive, the patient will be excluded from the protocol and referred for prenatal care.
* Being under oncological treatment (chemotherapy, radiotherapy and/or brachytherapy).
* Being on their period.
* Have a previous confirmatory diagnosis of HIV and/or hepatitis infection.
* Having taken antiplatelet medications, e.g., acetylsalicylic acid, at least 24 hours before the study.

Discontinuation Criteria:

* If the participant refuses any of the study procedures.
* If the study gynecologist detects that the participant has had a hysterectomy.
* If the volume of the biological samples is insufficient (less than 10 mL for the blood sample).

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Liquid-based Cytology LBC results (categorical) | Cervical smear will be taken during the first visit (Day 1). LBC results will be available within a maximum of 20 days after sampling. This test will be performed by a Licensed Clinical laboratory. All participants will be subjected to this test.
  Study of cells -of the cervix- using a microscope. Cytology is the official screening test for cervical precursor lesions and/or cervical cancer in most countries.
  Cytology's results:
  Negative to lesion/malignancy. Negative with inflammation. Negative with sexually transmitted infection. Negative with HPV/Herpes cytopathic changes. Negative with atrophy. Positive with ASC-US. Positive with ASC-H. Positive with AGUS. Positive with CIN-1. Positive with CIN-2. Positive with CIN-3. Positive with carcinoma in situ. Positive with LSIL/HSIL. Positive with adenocarcinoma. Positive with Cancer/Malignancy. Positive with probable lesion/cancer/malignancy.
Molecular screening results (dichotomic) | Blood samples will be taken during the first visit (Day 1). Molecular screening results will be available within a maximum of 20 days after sampling. All participants will be subjected to this test.
  Molecular screening detects three human protein biomarkers in human sera by Western blot and ELISA. Western blot results are qualitative (band intensity units or IU) and ELISA results are quantitative (ng/mL). The final result for molecular screening test is computed as follows:
  Negative. Only if the three independent biomarkers are below their cutoff values.
  Positive. If any of the three independent biomarkers is equal to or greater than its cutoff value.
  Cutoff values are as follows:
  Biomarker 1 positive >= 1.37 IU. Biomarker 1 negative < 1.37 IU. Biomarker 2 positive >= 17.74 ng/mL. Biomarker 2 negative < 17.74 ng/mL. Biomarker 3 positive >= 0.38 IU. Biomarker 3 negative < 0.38 IU.
HPV test results (categorical) | Cervical smear will be taken during the first visit (Day 1). HPV test results will be available within a maximum of 20 days after sampling. This test will be performed by a Licensed Clinical laboratory. All participants will be subjected to this test.
  HPV test will detect fifteen different high-risk genotypes by PCR:
  HPV-16 genotype. HPV-18 genotype. HPV-pool (including HPV-31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 67, and 68 genotypes).
  The final test result will be assigned as follows:
  Positive HPV test: If at least one of the fifteen genotypes is detected. Negative HPV test: Only if none of the fifteen genotypes are detected.
Colposcopy diagnosis (categorical) | Colposcopy will be performed during the first visit (Day 1). This diagnostic test will be performed by a licensed gynecologist. All participants will be subjected to this diagnostic test. Colposcopy will be used as a reference test.
  Colposcopy is the exploration of the female genitalia -vulva, vagina, and cervix- using a lighted magnifying instrument (colposcope). Its accuracy is higher than that of the cytology. If the gynecologist detects/suspects a lesion or malignancy during colposcopy, a biopsy will be drawn for histopathologic analysis.
  Colposcopy results:
  Negative with no alterations. Negative with inflammation. Negative with condyloma/condylomatosis/HPV. Negative with atrophy. Negative with squamous metaplasia. Negative with ectropion/ectopy/cervical erosion/cervical eversion/glandular eversion.
  Negative with Nabothian cysts. Negative with cervical polyp. Negative with Lichen sclerosus. Positive with CIN-1. Positive with CIN-2. Positive with CIN-3. Positive with carcinoma in situ CIN-3. Positive with neoplasia/invasive neoplasia. Positive with LSIL/HSIL. Positive with probable lesion/CIN/LSIL/HSIL.
Histopathology diagnosis (cathegorical) | The biopsy for histopathology will be drawn during the first visit (Day 1). Biopsies will be drawn only from women with positive colposcopy results. Histopathology is the gold standard for cervical cancer diagnosis.
  Histopathology is the microscopic analysis of a stained slide of a cervical biopsy by a licensed pathologist. The standard staining is H&E (hematoxylin and eosin).
  Histopathology results:
  Negative with normal tissue. Negative with cervicitis. Negative with HPV/Herpes infection. Positive with CIN-1. Positive with CIN-2. Positive with CIN-3. Positive with carcinoma in situ CIN-3. Positive LSIL/HSIL. Positive with microinvasive/invasive cancer. Positive with adenocarcinoma. Positive with sarcoma and other tumors. Positive with carcinoma of unknown primary origin/unspecified malignancy.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | During the first visit (Day 1).
  The study physician will record the participants:
  Weight in kilograms (kg). Height in meters (m). The Body Mass Index will be calculated as follows: BMI = kg/m^2.
Blood pressure | During the first visit (Day 1).
  Blood pressure is the amount of force the blood uses to get through the circulatory system measured in mmHg. It consists of two measurements:
  Systolic pressure in mmHg, e.g., 120 mmHg. Diastolic pressure in mmHg, e.g., 80 mmHg. The final result will display the two independent measurements, e.g., 120/80 mmHg.
Ethnicity | During the first visit (Day 1) by clinical interview.
  Ethnicity data will be obtained through clinical interview. Ethnicity is linked to cultural expression and identity.
  Ethnicity options:
  Hispanic/Latino. Not Hispanic/Latino.
Race | During the first visit (Day 1) by clinical interview.
  Race data will be obtained through clinical interview. Race is linked to physical characteristics.
  Race options:
  American Indian. Alaska Native. Asian. Black or African American. African Mexican. Native Hawaiian or Other Pacific Islander. Mexican Original People. White.
Age at Menarche | During the first visit (Day 1) by clinical interview.
  Age at menarche -in years- will be obtained during the clinical interview. Menarche is the first menstrual period in a female adolescent, typically occurs between the ages of 10 and 16.
Age at sexual debut | During the first visit (Day 1) by clinical interview.
  The age at sexual debut -in years- will be obtained during the clinical interview. The age will be recorded in years.
Number of years since menarche to sexual debut | During the first visit (Day 1) by clinical interview.
  The number of years since menarche to sexual debut will be calculated as follows:
  NYSMSD = Age of Sexual Debut - Age of Menarche
Number of lifetime sexual partners | During the first visit (Day 1) by clinical interview.
  The number of lifetime sexual partners of the participants will be obtained during the clinical interview.
Number of years since last cytology | During the first visit (Day 1) by clinical interview.
  The year of last or previous cytology will be obtained during the clinical interview. The number of years since las cytology will be calculated as follows:
  NYSLCy =Year of Participation in the Study - Year of Last/Previous Cytology.
Number of years since colposcopy | During the first visit (Day 1) by clinical interview.
  The year of last or previous colposcopy will be obtained during the clinical interview. The number of years since last colposcopy will be calculated as follows:
  NYSLCo =Year of Participation in the Study - Year of Last/Previous Colposcopy.
Number of abortions | During the first visit (Day 1) by clinical interview.
  The number of abortions will be obtained during the clinical interview.
Number of vaginal deliveries | During the first visit (Day 1) by clinical interview.
  The number of vaginal deliveries will be obtained during the clinical interview
Number of Caesarean sections | During the first visit (Day 1) by clinical interview.
  The number of Caesarean sections will be obtained during the clinical interview.
Number of cigarettes per week | During the first visit (Day 1) by clinical interview.
  The number of cigarettes per week will be obtained during the clinical interview.

OTHER OUTCOMES:
p16 immunohistochemistry results (dichotomic) | This test will be performed using the remaining tissue from randomly selected biopsies. None of the participants will be biopsied more than once. Biopsies will be drawn during the first visit (Day 1) only if a lesion/malignancy is detected in colposcopy.
  This test detects the human biomarker p16INK4a widely used for assessing HPV infection in a cervical biopsy.
  P16 IHC results:
  Positive. Negative. Inconclusive.

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo E Gatica-Galina, MD in OB/GY & Gynecol Oncol, Principal Investigator — Clinica Reina Madre Metepec
Locations (1):
- Clinica Reina Madre Metepec, San Mateo Atenco, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No
All de-identified individual participant data will be publicly available in the supplementary material associated with the scientific publication.

REFERENCES:
- [Background] Serdar CC, Cihan M, Yucel D, Serdar MA. Sample size, power and effect size revisited: simplified and practical approaches in pre-clinical, clinical and laboratory studies. Biochem Med (Zagreb). 2021 Feb 15;31(1):010502. doi: 10.11613/BM.2021.010502. Epub 2020 Dec 15. PMID 33380887
- [Background] Rozemeijer K, Penning C, Siebers AG, Naber SK, Matthijsse SM, van Ballegooijen M, van Kemenade FJ, de Kok IM. Comparing SurePath, ThinPrep, and conventional cytology as primary test method: SurePath is associated with increased CIN II+ detection rates. Cancer Causes Control. 2016 Jan;27(1):15-25. doi: 10.1007/s10552-015-0678-1. Epub 2015 Oct 12. PMID 26458884
- [Background] Bell ML, Kenward MG, Fairclough DL, Horton NJ. Differential dropout and bias in randomised controlled trials: when it matters and when it may not. BMJ. 2013 Jan 21;346:e8668. doi: 10.1136/bmj.e8668. PMID 23338004
- [Background] Hajian-Tilaki K. Sample size estimation in diagnostic test studies of biomedical informatics. J Biomed Inform. 2014 Apr;48:193-204. doi: 10.1016/j.jbi.2014.02.013. Epub 2014 Feb 26. PMID 24582925
- [Background] DeLong ER, DeLong DM, Clarke-Pearson DL. Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach. Biometrics. 1988 Sep;44(3):837-45. PMID 3203132
- [Background] Hu ZY, Xiao L, Bode AM, Dong Z, Cao Y. Glycolytic genes in cancer cells are more than glucose metabolic regulators. J Mol Med (Berl). 2014 Aug;92(8):837-45. doi: 10.1007/s00109-014-1174-x. Epub 2014 Jun 8. PMID 24906457
- [Background] Xue C, Gu X, Li G, Bao Z, Li L. Expression and Functional Roles of Eukaryotic Initiation Factor 4A Family Proteins in Human Cancers. Front Cell Dev Biol. 2021 Nov 19;9:711965. doi: 10.3389/fcell.2021.711965. eCollection 2021. PMID 34869305
- [Background] Li H, Liu J, Shen S, Dai D, Cheng S, Dong X, Sun L, Guo X. Pan-cancer analysis of alternative splicing regulator heterogeneous nuclear ribonucleoproteins (hnRNPs) family and their prognostic potential. J Cell Mol Med. 2020 Oct;24(19):11111-11119. doi: 10.1111/jcmm.15558. Epub 2020 Sep 11. PMID 32915499
- [Background] Dreyfuss G, Matunis MJ, Pinol-Roma S, Burd CG. hnRNP proteins and the biogenesis of mRNA. Annu Rev Biochem. 1993;62:289-321. doi: 10.1146/annurev.bi.62.070193.001445. No abstract available. PMID 8352591
- [Background] Checa-Rojas A, Delgadillo-Silva LF, Velasco-Herrera MDC, Andrade-Dominguez A, Gil J, Santillan O, Lozano L, Toledo-Leyva A, Ramirez-Torres A, Talamas-Rohana P, Encarnacion-Guevara S. GSTM3 and GSTP1: novel players driving tumor progression in cervical cancer. Oncotarget. 2018 Apr 24;9(31):21696-21714. doi: 10.18632/oncotarget.24796. eCollection 2018 Apr 24. PMID 29774096
- [Background] William W, Ware A, Basaza-Ejiri AH, Obungoloch J. A pap-smear analysis tool (PAT) for detection of cervical cancer from pap-smear images. Biomed Eng Online. 2019 Feb 12;18(1):16. doi: 10.1186/s12938-019-0634-5. PMID 30755214
- [Background] Shin MB, Garcia PJ, Saldarriaga EM, Fiestas JL, Asbjornsdottir KH, Iribarren SJ, Barnabas RV, Gimbel S. Cost of community-based human papillomavirus self-sampling in Peru: A micro-costing study. Lancet Reg Health Am. 2022 Apr;8:100160. doi: 10.1016/j.lana.2021.100160. Epub 2021 Dec 29. PMID 35528707
- [Background] Giannella L, Di Giuseppe J, Delli Carpini G, Grelloni C, Fichera M, Sartini G, Caimmi S, Natalini L, Ciavattini A. HPV-Negative Adenocarcinomas of the Uterine Cervix: From Molecular Characterization to Clinical Implications. Int J Mol Sci. 2022 Nov 30;23(23):15022. doi: 10.3390/ijms232315022. PMID 36499345
- [Background] Jenkins D, Molijn A, Kazem S, Pirog EC, Alemany L, de Sanjose S, Dinjens W, Quint W. Molecular and pathological basis of HPV-negative cervical adenocarcinoma seen in a global study. Int J Cancer. 2020 Nov 1;147(9):2526-2536. doi: 10.1002/ijc.33124. Epub 2020 Jul 6. PMID 32474915
- [Background] Lee JE, Chung Y, Rhee S, Kim TH. Untold story of human cervical cancers: HPV-negative cervical cancer. BMB Rep. 2022 Sep;55(9):429-438. doi: 10.5483/BMBRep.2022.55.9.042. PMID 35725012
- [Background] Najib FS, Hashemi M, Shiravani Z, Poordast T, Sharifi S, Askary E. Diagnostic Accuracy of Cervical Pap Smear and Colposcopy in Detecting Premalignant and Malignant Lesions of Cervix. Indian J Surg Oncol. 2020 Sep;11(3):453-458. doi: 10.1007/s13193-020-01118-2. Epub 2020 Jun 23. PMID 33013127
- [Background] Mayrand MH, Duarte-Franco E, Rodrigues I, Walter SD, Hanley J, Ferenczy A, Ratnam S, Coutlee F, Franco EL; Canadian Cervical Cancer Screening Trial Study Group. Human papillomavirus DNA versus Papanicolaou screening tests for cervical cancer. N Engl J Med. 2007 Oct 18;357(16):1579-88. doi: 10.1056/NEJMoa071430. PMID 17942871
- [Background] Kitchener HC, Castle PE, Cox JT. Chapter 7: Achievements and limitations of cervical cytology screening. Vaccine. 2006 Aug 31;24 Suppl 3:S3/63-70. doi: 10.1016/j.vaccine.2006.05.113. PMID 16950019
- [Background] Bravington A, Chen H, Dyson J, Jones L, Dalgliesh C, Bryan A, Patnick J, Macleod U. Challenges and opportunities for cervical screening in women over the age of 50 years: a qualitative study. Br J Gen Pract. 2022 Nov 24;72(725):e873-e881. doi: 10.3399/BJGP.2022.0036. Print 2022 Dec. PMID 36192359
- [Background] Shin HY, Song SY, Jun JK, Kim KY, Kang P. Barriers and strategies for cervical cancer screening: What do female university students know and want? PLoS One. 2021 Oct 5;16(10):e0257529. doi: 10.1371/journal.pone.0257529. eCollection 2021. PMID 34610022
- [Background] Petersen Z, Jaca A, Ginindza TG, Maseko G, Takatshana S, Ndlovu P, Zondi N, Zungu N, Varghese C, Hunting G, Parham G, Simelela P, Moyo S. Barriers to uptake of cervical cancer screening services in low-and-middle-income countries: a systematic review. BMC Womens Health. 2022 Dec 2;22(1):486. doi: 10.1186/s12905-022-02043-y. PMID 36461001
- [Background] Akinlotan M, Bolin JN, Helduser J, Ojinnaka C, Lichorad A, McClellan D. Cervical Cancer Screening Barriers and Risk Factor Knowledge Among Uninsured Women. J Community Health. 2017 Aug;42(4):770-778. doi: 10.1007/s10900-017-0316-9. PMID 28155005
- [Background] Zhang L, Mosquera I, Lucas E, Rol ML, Carvalho AL, Basu P; CanScreen5 collaborators. CanScreen5, a global repository for breast, cervical and colorectal cancer screening programs. Nat Med. 2023 May;29(5):1135-1145. doi: 10.1038/s41591-023-02315-6. Epub 2023 Apr 27. PMID 37106168
- [Background] Mitra A, Tzafetas M, Lyons D, Fotopoulou C, Paraskevaidis E, Kyrgiou M. Cervical intraepithelial neoplasia: screening and management. Br J Hosp Med (Lond). 2016 Aug 2;77(8):C118-23. doi: 10.12968/hmed.2016.77.8.C118. No abstract available. PMID 27487071
- [Background] Alimena S, Davis J, Fichorova RN, Feldman S. The vaginal microbiome: A complex milieu affecting risk of human papillomavirus persistence and cervical cancer. Curr Probl Cancer. 2022 Aug;46(4):100877. doi: 10.1016/j.currproblcancer.2022.100877. Epub 2022 Jun 9. PMID 35709613
- [Background] Johnson CA, James D, Marzan A, Armaos M. Cervical Cancer: An Overview of Pathophysiology and Management. Semin Oncol Nurs. 2019 Apr;35(2):166-174. doi: 10.1016/j.soncn.2019.02.003. Epub 2019 Mar 14. PMID 30878194
- [Background] Ribeiro AA, Costa MC, Alves RR, Villa LL, Saddi VA, Carneiro MA, Zeferino LC, Rabelo-Santos SH. HPV infection and cervical neoplasia: associated risk factors. Infect Agent Cancer. 2015 May 26;10:16. doi: 10.1186/s13027-015-0011-3. eCollection 2015. PMID 26244052
- [Background] Vesco KK, Whitlock EP, Eder M, Burda BU, Senger CA, Lutz K. Risk factors and other epidemiologic considerations for cervical cancer screening: a narrative review for the U.S. Preventive Services Task Force. Ann Intern Med. 2011 Nov 15;155(10):698-705, W216. doi: 10.7326/0003-4819-155-10-201111150-00377. Epub 2011 Oct 17. PMID 22006929
- [Background] International Collaboration of Epidemiological Studies of Cervical Cancer. Cervical carcinoma and sexual behavior: collaborative reanalysis of individual data on 15,461 women with cervical carcinoma and 29,164 women without cervical carcinoma from 21 epidemiological studies. Cancer Epidemiol Biomarkers Prev. 2009 Apr;18(4):1060-9. doi: 10.1158/1055-9965.EPI-08-1186. Epub 2009 Mar 31. PMID 19336546
- [Background] Plummer M, Herrero R, Franceschi S, Meijer CJ, Snijders P, Bosch FX, de Sanjose S, Munoz N; IARC Multi-centre Cervical Cancer Study Group. Smoking and cervical cancer: pooled analysis of the IARC multi-centric case--control study. Cancer Causes Control. 2003 Nov;14(9):805-14. doi: 10.1023/b:caco.0000003811.98261.3e. PMID 14682438
- [Background] Collins S, Rollason TP, Young LS, Woodman CB. Cigarette smoking is an independent risk factor for cervical intraepithelial neoplasia in young women: a longitudinal study. Eur J Cancer. 2010 Jan;46(2):405-11. doi: 10.1016/j.ejca.2009.09.015. Epub 2009 Oct 12. PMID 19819687
- [Background] Tekalegn Y, Sahiledengle B, Woldeyohannes D, Atlaw D, Degno S, Desta F, Bekele K, Aseffa T, Gezahegn H, Kene C. High parity is associated with increased risk of cervical cancer: Systematic review and meta-analysis of case-control studies. Womens Health (Lond). 2022 Jan-Dec;18:17455065221075904. doi: 10.1177/17455065221075904. PMID 35114865
- [Background] Bezabih M, Tessema F, Sengi H, Deribew A. Risk Factors Associated with Invasive Cervical Carcinoma among Women Attending Jimma University Specialized Hospital, Southwest Ethiopia: A Case Control Study. Ethiop J Health Sci. 2015 Oct;25(4):345-52. doi: 10.4314/ejhs.v25i4.8. PMID 26949299
- [Background] McGraw SL, Ferrante JM. Update on prevention and screening of cervical cancer. World J Clin Oncol. 2014 Oct 10;5(4):744-52. doi: 10.5306/wjco.v5.i4.744. PMID 25302174
- [Background] Hwang LY, Ma Y, Benningfield SM, Clayton L, Hanson EN, Jay J, Jonte J, Godwin de Medina C, Moscicki AB. Factors that influence the rate of epithelial maturation in the cervix in healthy young women. J Adolesc Health. 2009 Feb;44(2):103-110. doi: 10.1016/j.jadohealth.2008.10.006. PMID 19167657
- [Background] Ruiz AM, Ruiz JE, Gavilanes AV, Eriksson T, Lehtinen M, Perez G, Sings HL, James MK, Haupt RM; FUTURE I and II Study Group. Proximity of first sexual intercourse to menarche and risk of high-grade cervical disease. J Infect Dis. 2012 Dec 15;206(12):1887-96. doi: 10.1093/infdis/jis612. Epub 2012 Oct 12. PMID 23066159
- [Background] Mok, S. C., Wong, K. K., Lu, K. H., Munger, K. & Nagymanyoki, Z. Molecular basis of gynecologic diseases. in Essential Concepts in Molecular Pathology 409-424 (Elsevier, 2020). doi:10.1016/B978-0-12-813257-9.00023-1.
- See also: World Health Organization & International Agency for Research on Cancer. Global Cancer Observatory — https://gco.iarc.fr/today/home
- See also: World Health Organization. Global Strategy to Accelerate the Elimination of Cervical Cancer as a Public Health Problem — https://www.who.int/publications/i/item/9789240014107
- See also: Sellors JW & Sankaranarayanan R. An introduction to Cervical Intraepithelial Neoplasia (CIN). in Colposcopy and treatment of cervical intraepithelial neoplasia: a beginners manual — https://screening.iarc.fr/colpo.php
- See also: International Agency for Research on Cancer. CanScreen5. Cervical Cancer Screening Programme. Country Fact Sheet: Mexico — https://canscreen5.iarc.fr/?page=countryfactsheetcervix&q=MEX&rc=
- See also: Mexico's Ministry of Health. NOM-014-SSA2-1994. For Prevention, Detection, Diagnosis, Treatment, Control and Epidemiological Surveillance of Cervical Cancer — https://www.gob.mx/cms/uploads/attachment/file/10397/NOM-014-SSA2-1994.pdf
- See also: World Health Organization. WHO Guideline for Screening and Treatment of Cervical Pre-Cancer Lesions for Cervical Cancer Prevention. — https://www.who.int/publications/i/item/9789240030824
- See also: Mexican Social Security Institute (IMSS) & Mexican Government. Clinical Practice Guidelines. Prevention and Timely Detection of Cervical Cancer at the First-Level of Care — https://www.imss.gob.mx/sites/all/statics/guiasclinicas/146GER.pdf
- See also: William, W., Ware, A., Basaza-Ejiri, A. H. & Obungoloch, J. Automated diagnosis and classification of cervical cancer from Pap-smear images. in 2019 IST-Africa Week Conference, IST-Africa 2019 — https://ieeexplore.ieee.org/document/8764887
- See also: Reyes-Hernández, D. O. et al. Novel Serum Protein Biomarkers for Precancerous Cervical Lesions and Cervical Cancer. Glob J Health Sci 16, 44 (2024). — https://ccsenet.org/journal/index.php/gjhs/article/view/0/50473
- See also: Mexican Social Security Institute (IMSS) & Mexican Government. Clinical Practice Guidelines. Treatment of Cervical Cancer at the Second and Third-Level of Care — https://www.imss.gob.mx/sites/all/statics/guiasclinicas/333GER.pdf